CLINICAL TRIAL: NCT01000818
Title: An Open-Label, 3-Period, Fixed-Sequence Study to Evaluate the Effect of Famotidine and Omeprazole on MK0518 Pharmacokinetics in HIV-Infected Patients on a Stable MK0518-Containing Regimen
Brief Title: A Study to Evaluate the Effect of Famotidine and Omeprazole on MK0518 (Raltegravir) Pharmacokinetics in Human Immunodeficiency Virus (HIV)-Infected Patients (0518-054)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0518-054; MK0518-054; 2009_681
Record Dates: First submitted 2009-10-22; First posted 2009-10-23 (Estimated); Results first posted 2010-05-28 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-02

CONDITIONS: HIV-1 Infection; HIV Infections
Keywords: Treatment experienced
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium; Famotidine; Omeprazole

ARMS (3):
- Period 1 (Experimental): MK0518
  Interventions: Drug: MK0518 (Raltegravir)
- Period 2 (Experimental): famotidine + MK0518
  Interventions: Drug: MK0518 (Raltegravir); Drug: famotidine
- Period 3 (Experimental): omeprazole + MK0518
  Interventions: Drug: MK0518 (Raltegravir); Drug: omeprazole

INTERVENTIONS:
Drug: MK0518 (Raltegravir) — 400 mg oral tablet of MK0518 once every 12 hours. Period 1 duration is one day, Period 2 duration is one day, Period 3 duration is five days.
  Other Names: Raltegravir
Drug: famotidine — Single 20 mg famotidine oral tablet taken 2 hours prior to administration of AM dose of MK0518
  Arms: Period 2
Drug: omeprazole — 20 mg oral tablet of omeprazole, once daily for 5 days
  Arms: Period 3

SUMMARY:
An open-label, 3-period, fixed-sequence study in a panel of 18 HIV-infected patients on MK0518 as part of a stable treatment regimen for HIV.

ELIGIBILITY:
Inclusion Criteria:

* Patient is Human immunodeficiency virus (HIV) positive
* Patient is taking an MK0518 (Raltegravir) containing regimen
* Patient has not had any changes to his/her antiviral regimen in the last 2 weeks
* Patient who is of reproductive potential agrees to use an acceptable method of birth control
* Patients baseline health is stable

Exclusion Criteria:

* Patient has a history of stroke or chronic seizures.
* Patient has a history of gastric bypass surgery
* Patient is pregnant of breastfeeding
* Patient consumes excessive amounts of caffeinated beverages daily
* Patient has had major surgery, donated blood, or participated in another investigational study in the past 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-06; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through Abbott Northwestern Hospital Infectious Diseases Clinic, Minneapolis, MN and Prism Research, St. Paul, MN, between June 2008 and March 2009.
Pre-assignment Details: A total of 18 participants were enrolled in the study.
Groups:
- Raltegravir/Famotidine/Omeprazole: Period 1 - 400 mg Raltegravir x 1 day
  Period 2 - 20 mg Famotidine + 400 mg Raltegravir x 1 day
  Period 3 - 20 mg Omeprazole + 400 mg Raltegravir x 5 days
Period: Raltegravir
Arm/Group | Raltegravir/Famotidine/Omeprazole
Started | 18
Completed | 18
Not Completed | 0
Period: Famotidine + Raltegravir
Arm/Group | Raltegravir/Famotidine/Omeprazole
Started | 18
Completed | 18
Not Completed | 0
Period: Omeprazole + Raltegravir
Arm/Group | Raltegravir/Famotidine/Omeprazole
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Raltegravir/Famotidine/Omeprazole
Number analyzed (Participants) | 18
Age, Continuous [Mean (Full Range); unit: years] | 49.3 [37 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 16
Height [Mean (Full Range); unit: Centimeters] | 176.6 [161.0 to 188.0]
Weight [Mean (Full Range); unit: Kilograms] | 85.7 [60.6 to 141.0]

OUTCOME MEASURES:

1. Primary Outcome: Plasma Area Under Curve (AUC 0-12 hr ) for Raltegravir
Description: Area Under the Plasma Concentration-Time Curve and peak concentration
Time Frame: 12 hours postdose
Population: Eighteen HIV-Infected Patients
Measure: Geometric Mean (95% Confidence Interval); unit: µM*hr
Groups:
- 400 mg Raltegravir: Period 1 - 400 mg Raltegravir
- 20 mg Famotidine + 400 mg Raltegravir: Period 2 - 20 mg Famotidine + 400 mg Raltegravir
- 20 mg Omeprazole + 400 mg Raltegravir: Period 3 - 20 mg Omeprazole + 400 mg Raltegravir x 5days
Arm/Group | 400 mg Raltegravir | 20 mg Famotidine + 400 mg Raltegravir | 20 mg Omeprazole + 400 mg Raltegravir
Number analyzed (Participants) | 18 | 18 | 18
µM*hr | 12.36 [8.96 to 17.04] | 17.95 [13.02 to 24.75] | 17.12 [12.42 to 23.61]
Statistical Analysis 1: Comparison: 400 mg Raltegravir vs 20 mg Omeprazole + 400 mg Raltegravir; Test type: Non-Inferiority or Equivalence — The raltegravir AUC0-12 hr geometric mean ratio (raltegravir + omeprazole/raltegravir) is noniferior at less than 2.0; Geometric Mean Ratio = 1.39, 95% CI [1.04 to 1.84]
Statistical Analysis 2: Comparison: 400 mg Raltegravir vs 20 mg Famotidine + 400 mg Raltegravir; Test type: Non-Inferiority or Equivalence — The raltegravir AUC0-12 hr geometric mean ratio (raltegravir + omeprazole/raltegravir) is noniferior at less than 2.0; Geometric Mean Ratio = 1.45, 95% CI [1.09 to 1.93]

ADVERSE EVENTS:
Arm/Group | Prestudy | 400 mg Raltegravir | 20 mg Famotidine + 400 mg Raltegravir | 20 mg Omeprazole + 400 mg Raltegravir
Serious Adverse Events (participants affected / at risk) | 1/18 | 0/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 2/18 | 1/18 | 6/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prestudy (N=18) | 400 mg Raltegravir (N=18) | 20 mg Famotidine + 400 mg Raltegravir (N=18) | 20 mg Omeprazole + 400 mg Raltegravir (N=18)
Ruptured coronary artery plaque (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prestudy (N=18) | 400 mg Raltegravir (N=18) | 20 mg Famotidine + 400 mg Raltegravir (N=18) | 20 mg Omeprazole + 400 mg Raltegravir (N=18)
Abnormal feces (Gastrointestinal disorders) | 0 (0) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 (0) | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 | 0 | 1
vomiting (Gastrointestinal disorders) | 0 (0) | 2 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 | 0 | 1
Knee pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 (0) | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication guidelines.